CLINICAL TRIAL: NCT04397406
Title: Role of Dexmedetomidine or Fentanyl as Additives to Epidural Levobupivacaine in Painless Labor: A Double Blind Randomized Controlled Study
Brief Title: Dexmedetomidine or Fentanyl as Additives to Epidural Levobupivacaine in Painless Labor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hend Mahmoud Moneeb El-shazly, Assistant lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 33447/10/19
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Epidural Analgesia; Painless Labor; Dexmedetomidine; Fentanyl; Levobupivacaine
MeSH Terms: interventions — Levobupivacaine; Dexmedetomidine; Fentanyl

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated into three equal groups by computer generated sequence through sealed opaque envelopes. Each group will include 30 patients.
  Group C (Control group): Epidural analgesia with levobupivacaine alone Group D (Dexmedetomidine group): Epidural analgesia with levobupivacaine and dexmedetomidine Group F (Fentanyl group): Epidural analgesia with levobupivacaine and fentanyl
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group C (Control group) (Active Comparator): pidural analgesia with levobupivacaine alone
  Interventions: Drug: levobupivacaine
- Group D (Dexmedetomidine group) (Experimental): Epidural analgesia with levobupivacaine and dexmedetomidine
  Interventions: Drug: levobupivacaine; Drug: Dexmedetomidine
- Group F (Fentanyl group) (Experimental): Epidural analgesia with levobupivacaine and fentanyl
  Interventions: Drug: levobupivacaine; Drug: Fentanyl

INTERVENTIONS:
Drug: levobupivacaine — The patients will receive 15 ml of 0.125% levobupivacaine.
Drug: Dexmedetomidine — The patients will receive 13 ml of 0.125% levobupivacaine and 0.5μg/kg dexmedetomidine diluted in 2 ml saline.
  Arms: Group D (Dexmedetomidine group)
Drug: Fentanyl — The patients will receive 13 ml of 0.125% levobupivacaine and 25μg fentanyl diluted in 2 ml saline.
  Arms: Group F (Fentanyl group)

SUMMARY:
Central neuraxial analgesia has been extensively used for labor analgesia and is currently the gold standard technique for pain control in obstetrics.

The aim of the study will be to compare the role of dexmedetomidine or fentanyl as additives to epidural levobupivacaine in painless vaginal delivery as regard maternal analgesia and safety.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status class II and III,
* Full term pregnancy.

Exclusion Criteria:

* Patient refusal to epidural analgesia,
* Contraindications of epidural analgesia (coagulopathy, local infection, vertebral deformity hypersensitivity to levobupivacaine, dexmedetomidine or fentanyl, hemodynamic instability, severe aortic or mitral stenosis),
* Cardiac diseases
* Severe pre-eclampsia,
* Breech presentations
* Antepartum hemorrhage
* Cephalopelvic disproportion
* Body mass index ≥40 kg/m2.

Ages: 21 Years to 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Duration of maternal analgesia | 24 hours after epidural injection
  Duration of analgesia will be assessed by measuring the time between the onset of sensory block and return of pain sensation. If the block is inadequate or the patient has pain, a top up dose of 8 mL of the study medication and local anesthetic will be given when visual analogue scale (VAS) will be ≥ 4.
  The pain relief will be assessed by the visual analogue scale (VAS) from 0 to 10 (0: no pain, 1-3: mild pain, 4-7: moderate pain, > 7: severe pain).

SECONDARY OUTCOMES:
Onset of maternal analgesia. | One hour after epidural injection
  The onset of analgesia will be defined as the time taken from drug administration to visual analogue scale (VAS) <3.
Complications of drugs of epidural technique | 24 hours after epidural injection
  Drugs: Sedation, Bradycardia Epidural anesthesia (including nausea, vomiting, backache and fever)

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No